CLINICAL TRIAL: NCT03804853
Title: Immediate Accelerated Shoulder Rehabilitation Versus a Standard Protocol Following Reverse Total Shoulder Arthroplasty: A Randomized Controlled Trial
Brief Title: Rehabilitation Following Reverse Total Shoulder Arthroplasty
Acronym: RTSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: TRIA Orthopaedic Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-259
Record Dates: First submitted 2019-01-08; First posted 2019-01-15 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Shoulder Osteoarthritis
Keywords: Rehabilitiation; Reverse total shoulder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Active Shoulder Rehabilitation (Experimental)
  Interventions: Other: Rehabilitiation
- Traditional Should Rehabilitation (Active Comparator)
  Interventions: Other: Rehabilitiation

INTERVENTIONS:
Other: Rehabilitiation — This study will be a non-blinded randomized controlled outcomes study evaluating outcomes at baseline, 2 weeks, 6 weeks, 3 months, 6 months, and 1 year post-operatively from a primary reverse total shoulder arthroplasty with two different post-operative physical rehabilitation protocols. There will be 2 groups, one undergoing the immediate active shoulder physical therapy protocol consisting of four quadrant stretches and full active motion of the shoulder from post op day 1 in the hospital. The second group will follow the traditional TRIA physical therapy protocol consisting of PT (standard of care) followed by a gradual return to active range of motion of the shoulder beginning by week 6, calling for 18 physical therapy visits. The physical therapy will occur where the patient is most comfortable receiving it.

SUMMARY:
Reverse total shoulder arthroplasty (RTSA) has been successful in patients with rotator cuff arthropathy, proximal humerus fractures, failed primary total shoulder arthroplasty or failed hemiarthroplasty, and massive irreparable rotator cuff tear. Patients who undergo an RTSA report pain relief and functional range of motion. It has been more than 20 years since the advent of the RTSA construct but an immediate post-operative rehabilitation with active shoulder range of motion has not been prospectively studied in comparison to the traditional post-operative rehabilitation highlighted by Boudreau et al.12 Investigators plan to prospectively follow our patients following RTSA undergoing an immediate active shoulder rehabilitation (IASR) vs traditional rehabilitation in a randomized controlled fashion. Investigators plan to document clinical outcomes, complications and cost effectiveness out to 1 year.

The study will hopefully fulfill the Triple Aim model for HealthPartners by improving the health of the population, improve the experience of each individual, and make healthcare affordable by decreasing the total cost of care.

ELIGIBILITY:
Inclusion Criteria:

* > 55 years of age.
* Candidate for a primary reverse total shoulder arthroplasty.
* Capable of completing self-administered questionnaires.
* Be willing and able to return for all study-related follow-up procedures.
* Able and willing to give informed consent.
* Proficient in the English language.

Exclusion Criteria:

In-Clinic:

* Patients planning on undergoing a Primary Reverse Shoulder Total Arthroplasty due to proximal humeral fracture.
* Previous shoulder surgery including previous total shoulder arthroplasty or reverse total shoulder arthroplasty or hemiarthroplasty, or instability repairs
* Active bacterial infection of the shoulder.
* Any concomitant shoulder procedure.
* Additional ipsilateral or contralateral upper limb pathology that requires active treatment (i.e. surgery or brace).
* Inflammatory arthropathy.
* Diagnosed with Rheumatoid arthritis
* Diagnosed with gout.
* Subject is on chronic anticoagulation due to a bleeding disorder or has taken anticoagulants within 10 days prior to surgery.
* Peripheral vascular disease or other vascular disorders that would impair healing.
* Peripheral neuropathy or other neurological disorders that may impair the patient to ambulate.
* Patient is on workers compensation.
* Any condition requiring chemotherapy.
* Active tobacco user or former tobacco user who is not free of using tobacco for 8 weeks.
* Uncontrolled Diabetes Mellitus with an HbA1C > 7.5%.
* Current drug or alcohol abuse.
* Major medical illness (life expectancy less then 2 years or unacceptably high operative risk)
* Suspicion of cervical radiculopathy or myelopathy.
* Deltoid insufficiency on physical examination.

Intra-operative:

• Iatrogenic glenoid fracture

Post-operative:

* Neurological injury of the upper extremity.
* Complications from Primary Reverse Shoulder Total Arthroplasty (i.e. post-operative infection, bleeding, hardware failure).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
American Society for Elbow and Shoulder Score | Pre-operatively
  1. American Shoulder and Elbow score (ASES) is a scale that measures shoulder pain and function with 11 items, one item for pain and 10 items for function. The score for each subscale is out of 50 (0-50), with a higher score indicating a better outcome. The total score is a sum of both subscales, ranging between 0-100, using the following formula, Total score = ((10 - VAS pain) × 5) + (5/3 × sum of function items).
American Society for Elbow and Shoulder Score | 2 weeks
  1. American Shoulder and Elbow score (ASES) is a scale that measures shoulder pain and function with 11 items, one item for pain and 10 items for function. The score for each subscale is out of 50 (0-50), with a higher score indicating a better outcome. The total score is a sum of both subscales, ranging between 0-100, using the following formula, Total score = ((10 - VAS pain) × 5) + (5/3 × sum of function items).
American Society for Elbow and Shoulder Score | 3 months
  1. American Shoulder and Elbow score (ASES) is a scale that measures shoulder pain and function with 11 items, one item for pain and 10 items for function. The score for each subscale is out of 50 (0-50), with a higher score indicating a better outcome. The total score is a sum of both subscales, ranging between 0-100, using the following formula, Total score = ((10 - VAS pain) × 5) + (5/3 × sum of function items).
American Society for Elbow and Shoulder Score | 6 months
  1. American Shoulder and Elbow score (ASES) is a scale that measures shoulder pain and function with 11 items, one item for pain and 10 items for function. The score for each subscale is out of 50 (0-50), with a higher score indicating a better outcome. The total score is a sum of both subscales, ranging between 0-100, using the following formula, Total score = ((10 - VAS pain) × 5) + (5/3 × sum of function items).
American Society for Elbow and Shoulder Score | 1 year
  1. American Shoulder and Elbow score (ASES) is a scale that measures shoulder pain and function with 11 items, one item for pain and 10 items for function. The score for each subscale is out of 50 (0-50), with a higher score indicating a better outcome. The total score is a sum of both subscales, ranging between 0-100, using the following formula, Total score = ((10 - VAS pain) × 5) + (5/3 × sum of function items).
Simple Shoulder Test | Pre-operatively
  2. The Simple Shoulder Test Score (SST) is a 12 item, yes/no questionnaire assessing shoulder function. There are 2 items on function related to pain, 7 items about functions/strength and 3 items about range of motion. There are no subscales. A "yes" response is 1 point and a "no" response is 0 point. The following formula is used to calculate a score out of 100 (0-100), total= number of "yes" items/number of completed items × 100 = % "yes" responses. A higher score indicates better function from a scale of 0-100.
Simple Shoulder Test | 2 weeks
  2. The Simple Shoulder Test Score (SST) is a 12 item, yes/no questionnaire assessing shoulder function. There are 2 items on function related to pain, 7 items about functions/strength and 3 items about range of motion. There are no subscales. A "yes" response is 1 point and a "no" response is 0 point. The following formula is used to calculate a score out of 100 (0-100), total= number of "yes" items/number of completed items × 100 = % "yes" responses. A higher score indicates better function from a scale of 0-100.
Simple Shoulder Test | 3 months
  2. The Simple Shoulder Test Score (SST) is a 12 item, yes/no questionnaire assessing shoulder function. There are 2 items on function related to pain, 7 items about functions/strength and 3 items about range of motion. There are no subscales. A "yes" response is 1 point and a "no" response is 0 point. The following formula is used to calculate a score out of 100 (0-100), total= number of "yes" items/number of completed items × 100 = % "yes" responses. A higher score indicates better function from a scale of 0-100.
Simple Shoulder Test | 6 months
  2. The Simple Shoulder Test Score (SST) is a 12 item, yes/no questionnaire assessing shoulder function. There are 2 items on function related to pain, 7 items about functions/strength and 3 items about range of motion. There are no subscales. A "yes" response is 1 point and a "no" response is 0 point. The following formula is used to calculate a score out of 100 (0-100), total= number of "yes" items/number of completed items × 100 = % "yes" responses. A higher score indicates better function from a scale of 0-100.
Simple Shoulder Test | 1 year
  2. The Simple Shoulder Test Score (SST) is a 12 item, yes/no questionnaire assessing shoulder function. There are 2 items on function related to pain, 7 items about functions/strength and 3 items about range of motion. There are no subscales. A "yes" response is 1 point and a "no" response is 0 point. The following formula is used to calculate a score out of 100 (0-100), total= number of "yes" items/number of completed items × 100 = % "yes" responses. A higher score indicates better function from a scale of 0-100.
PROMIS Global 10 | Pre-operatively
  3. The PROMIS Global-10 is a global health quality of life patient reported outcome tool. It is part of the Patient-Reported Outcomes Measurement Information System (PROMIS). It measures symptoms, functioning, and healthcare quality of life for a wide variety of conditions. The PROMIS Global-10 consists of 10 questions assessing physical health, mental health, social health, pain, fatigue, and overall perceived quality of life. 7 questions inquire about health in "general" and 3 questions assess emotional problems, fatigue and pain in the last 7 days. Raw subscale scores for physical and mental health each are calculated out of 20. The raw score are converted to T scores for physical and mental health using the following formulas: the Global Physical Health score is generated by summing responses to Global03, Global06, Global07rescored, and Global08rescored. The Global Mental Health score is generated by summing responses to Global02, Global04, Global05, and Global10rescored.
PROMIS Global 10 | 2 weeks
  3. The PROMIS Global-10 is a global health quality of life patient reported outcome tool. It is part of the Patient-Reported Outcomes Measurement Information System (PROMIS). It measures symptoms, functioning, and healthcare quality of life for a wide variety of conditions. The PROMIS Global-10 consists of 10 questions assessing physical health, mental health, social health, pain, fatigue, and overall perceived quality of life. 7 questions inquire about health in "general" and 3 questions assess emotional problems, fatigue and pain in the last 7 days. Raw subscale scores for physical and mental health each are calculated out of 20. The raw score are converted to T scores for physical and mental health using the following formulas: the Global Physical Health score is generated by summing responses to Global03, Global06, Global07rescored, and Global08rescored. The Global Mental Health score is generated by summing responses to Global02, Global04, Global05, and Global10rescored.
PROMIS Global 10 | 3 months
  3. The PROMIS Global-10 is a global health quality of life patient reported outcome tool. It is part of the Patient-Reported Outcomes Measurement Information System (PROMIS). It measures symptoms, functioning, and healthcare quality of life for a wide variety of conditions. The PROMIS Global-10 consists of 10 questions assessing physical health, mental health, social health, pain, fatigue, and overall perceived quality of life. 7 questions inquire about health in "general" and 3 questions assess emotional problems, fatigue and pain in the last 7 days. Raw subscale scores for physical and mental health each are calculated out of 20. The raw score are converted to T scores for physical and mental health using the following formulas: the Global Physical Health score is generated by summing responses to Global03, Global06, Global07rescored, and Global08rescored. The Global Mental Health score is generated by summing responses to Global02, Global04, Global05, and Global10rescored.
PROMIS Global 10 | 6 months
  3. The PROMIS Global-10 is a global health quality of life patient reported outcome tool. It is part of the Patient-Reported Outcomes Measurement Information System (PROMIS). It measures symptoms, functioning, and healthcare quality of life for a wide variety of conditions. The PROMIS Global-10 consists of 10 questions assessing physical health, mental health, social health, pain, fatigue, and overall perceived quality of life. 7 questions inquire about health in "general" and 3 questions assess emotional problems, fatigue and pain in the last 7 days. Raw subscale scores for physical and mental health each are calculated out of 20. The raw score are converted to T scores for physical and mental health using the following formulas: the Global Physical Health score is generated by summing responses to Global03, Global06, Global07rescored, and Global08rescored. The Global Mental Health score is generated by summing responses to Global02, Global04, Global05, and Global10rescored.
PROMIS Global 10 | 1 year
  3. The PROMIS Global-10 is a global health quality of life patient reported outcome tool. It is part of the Patient-Reported Outcomes Measurement Information System (PROMIS). It measures symptoms, functioning, and healthcare quality of life for a wide variety of conditions. The PROMIS Global-10 consists of 10 questions assessing physical health, mental health, social health, pain, fatigue, and overall perceived quality of life. 7 questions inquire about health in "general" and 3 questions assess emotional problems, fatigue and pain in the last 7 days. Raw subscale scores for physical and mental health each are calculated out of 20. The raw score are converted to T scores for physical and mental health using the following formulas: the Global Physical Health score is generated by summing responses to Global03, Global06, Global07rescored, and Global08rescored. The Global Mental Health score is generated by summing responses to Global02, Global04, Global05, and Global10rescored.
Range of Motion | Pre-operatively, 3 months, 6 months, 1 year post-operatively
  4. Range of motion (ROM) of the shoulder is an objective measure of shoulder function. A blinded examiner will measure the range of motion in forward elevation, external rotation in the neutral position external rotation with the arm in abduction, internal rotation in the neutral position, and internal rotation with the arm in abduction. A goniometer will be used measuring to the nearest degree. The range of motion for forward elevation will range between 0-180 degrees with a higher number indicating a better outcome. External and internal rotation ranges from 0-90 degrees with a higher number indicating a better outcome.
Range of Motion | 3 months
  4. Range of motion (ROM) of the shoulder is an objective measure of shoulder function. A blinded examiner will measure the range of motion in forward elevation, external rotation in the neutral position external rotation with the arm in abduction, internal rotation in the neutral position, and internal rotation with the arm in abduction. A goniometer will be used measuring to the nearest degree. The range of motion for forward elevation will range between 0-180 degrees with a higher number indicating a better outcome. External and internal rotation ranges from 0-90 degrees with a higher number indicating a better outcome.
Range of Motion | 6 months
  4. Range of motion (ROM) of the shoulder is an objective measure of shoulder function. A blinded examiner will measure the range of motion in forward elevation, external rotation in the neutral position external rotation with the arm in abduction, internal rotation in the neutral position, and internal rotation with the arm in abduction. A goniometer will be used measuring to the nearest degree. The range of motion for forward elevation will range between 0-180 degrees with a higher number indicating a better outcome. External and internal rotation ranges from 0-90 degrees with a higher number indicating a better outcome.
Range of Motion | 1 year
  4. Range of motion (ROM) of the shoulder is an objective measure of shoulder function. A blinded examiner will measure the range of motion in forward elevation, external rotation in the neutral position external rotation with the arm in abduction, internal rotation in the neutral position, and internal rotation with the arm in abduction. A goniometer will be used measuring to the nearest degree. The range of motion for forward elevation will range between 0-180 degrees with a higher number indicating a better outcome. External and internal rotation ranges from 0-90 degrees with a higher number indicating a better outcome.

SECONDARY OUTCOMES:
Subscapularis Tear | 1 year
  Determination if a tear is present.

OTHER OUTCOMES:
Number of PT Visits | 1 Year
  Count of number of visits.

CONTACTS AND LOCATIONS:
Locations (1):
- TRIA Orthopaedic Center, Bloomington, Minnesota, United States